CLINICAL TRIAL: NCT01919138
Title: Outcomes of Severe Sepsis Patients in Surgical Intensive Care Units of National Taiwan University Hospital: Retrospective Review
Brief Title: Outcomes of Severe Sepsis Patients in Surgical Intensive Care Units
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201305085RINC
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- severe sepsis, septic shock

SUMMARY:
Retrospective review of the outcomes of severe sepsis patients in Surgical Intensive Care Unit of National Taiwan University Hospital from January 1, 2009 to December 31, 2011.

DETAILED DESCRIPTION:
Patients suffered from severe sepsis or septic shock have a mortality of 20~54%. It is major healthcare problems, affecting millions of individuals around the world each year. An international group of experts in the diagnosis and management of infection and sepsis, representing 11 organizations, published the first internationally accepted guidelines that the bedside clinician could use to improve outcomes in severe sepsis and septic shock in 2004, and further outcome was reported in 2008. Lots of medical centers have joined the Surviving Sepsis Campaign and follow the latest guideline. Many reports have shown that Surviving Sepsis Campaign Guideline can reduce patient mortality.

In surgical intensive care units of National Taiwan University Hospital (NTUH), the Surviving Sepsis Campaign Guideline was conducted since 2009. Our purpose is to investigate the characteristics and outcomes of severe sepsis patient in surgical intensive care units of NTUH by retrospective review of medical chart.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed as severe sepsis in Surgical Intensive Care units of National Taiwan University Hospital

Exclusion Criteria:

* < 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paitent with Severe Spesis in Surgical Intensive Care Units of National Taiwan University Hospital
Sampling Method: Probability Sample
Enrollment: 762 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
survival rate of severe sepsis patients in Surgical Intensive Care Units | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, MD, PhD, Principal Investigator — Department of Anesthesiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan